CLINICAL TRIAL: NCT01201499
Title: The Impact of Two Different Intraoperative Analgesia Techniques on Post-operative Outcome After Hepato-pancreato-biliary Surgery
Brief Title: Comparing the Outcome of Two Intraoperative Analgesia Techniques After Hepato-pancreato-biliary Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Professor Idit Matot. Chair, Department of Anesthsiology & Intensive Care, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-10-IM-0073-CTIL
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Pain; Analgesia; Sedation
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrathecal morphine (Active Comparator): A single shot of intrathecal morphine given before the induction of general anesthesia. Followed by postoperative IV patient-controlled morphine analgesia.
  Interventions: Drug: Intrathecal morphine
- Continuous IV remifentanil (Active Comparator): Continuous administration of IV remifentanil during surgery, supported by a single bolus of IV morphine at the end of surgery. Followed by postoperative IV patient-controlled morphine analgesia.
  Interventions: Drug: Continuous IV remifentanil

INTERVENTIONS:
Drug: Intrathecal morphine — a single dose of intrathecal morphine (ITM, 4 µcg/kg, or ~0.1-0.3 mg morphine before induction of general anesthesia, followed by postoperative patient-controlled morphine analgesia (IV-PCA) for postoperative pain.
  Other Names: ITM
  Arms: Intrathecal morphine
Drug: Continuous IV remifentanil — a continuous infusion of IV remifentanil supported by a single bolus of IV morphine, 0.2 mg/kg at the end of surgery, followed by IV-PCA morphine.
  Other Names: IVR
  Arms: Continuous IV remifentanil

SUMMARY:
Inadequate pain control after abdominal procedures may lead to adverse postoperative outcome. Epidural analgesia is currently an accepted technique in abdominal surgery, but its use has been limited in liver resections by postoperative coagulation disturbances and the possible increased risk of bleeding complications, including spinal hematoma. A range of alternative analgesic techniques can be used for major liver or pancreatic resections, including intrathecal morphine (single shot) administered immediately before surgery, and continuous administration of intravenous (IV) short-acting opioids, such as remifentanil, plus a single bolus of IV morphine. Postoperatively analgesia may be obtained by patient-controlled morphine analgesia (IV PCA). Both protocols have been demonstrated to provide satisfactory postoperative pain relief, and each has its unique advantages. However, to this end there is no data in the literature to show benefit from one regimen over the other. We therefore wish to determine whether there is a difference in analgesic efficacy between the two techniques, as optimizing perioperative pain relief in this rapidly expanding surgical field is of utmost importance. Our hypothesis is that continuous intraoperative IV analgesia with remifentanil followed by IV PCA morphine is not inferior to intrathecal morphine with respect to analgesia and ambulation outcome, and may provide an alternative, non-invasive intraoperative analgesic technique.

DETAILED DESCRIPTION:
BACKGROUND Inadequate pain control after abdominal procedures might result in increased morbidity, length of stay, and delay in overall recovery. Epidural analgesia is currently an accepted technique in major abdominal surgery [1-4]. Postoperative coagulation disturbances related to liver surgery, even in patients with normal preoperative coagulation undergoing uncomplicated hepatectomy, raises concerns about the safety of postoperative analgesia administered through an epidural catheter. Coagulation changes after liver surgery and the possible increased risk of bleeding complications, including spinal hematoma, have limited the use of epidural analgesia [5-7].

A range of alternative analgesic techniques can be used for major liver or pancreatic resections. A single dose of intrathecal morphine (ITM), administered immediately before surgery, followed by postoperative patient-controlled morphine analgesia (IV PCA), has been demonstrated to provide satisfactory postoperative pain relief which was not inferior to continuous epidural analgesia up to 48 hours after hepatic surgery [8, 9]. Another study in patients undergoing hepato-pancreato-biliary surgery has shown that ITM, compared with thoracic epidural analgesia, is associated with a reduced incidence of postoperative hypotension, intravenous fluid requirements, hospitalization, and incidence of respiratory complications [10]. Alternatively, few reports have demonstrated the advantage of using continuous administration of intravenous (IV) short-acting opioids, such as remifentanil. This regime has been shown to facilitate earlier extubation, to provide excellent intraoperative hemodynamic stability and rapid recovery [11]. Nevertheless, as remifentanil is rapidly metabolized, there is a need at the end of surgery to initiate another post-operative pain strategy to prevent unacceptable pain in the post-operative period. This has been accomplished by the administration of morphine which has been shown to provide an effective postoperative pain control (a bolus followed by IV PCA).

To date, these two analgesic regimens (ITM vs. continuous IV remifentanil) are frequently used in our institution. Nevertheless, there is no data in the literature to show benefit from one regimen over the other. We therefore wish to determine whether there is a difference in analgesic efficacy between the two techniques as optimizing perioperative pain relief in this rapidly expanding surgical field is of utmost importance.

METHODS Study design The study will be conducted as a prospective, randomized, double blinded one. Intra-operatively, anesthesia and surgical management will follow the routines. Intravenous fluid and blood supplements will be administered according to the anesthesiologists' decision. Also, the decision to extubate the patient at the end of surgery will be left to the discretion of the anesthesiologist. Post-operatively, all patients will be transferred to the ICU or to the recovery room for at least 24 hours. Patients may also be transferred first to the recovery room and than to the ICU. These are the routines in our hospital.

Consented patients will be randomly allocated to two groups by a computer-generated list:

Group 1 will receive a single dose of intrathecal morphine (ITM, 4 µcg/kg, or ~0.1-0.3 mg morphine)[10, 12-14] before induction of general anesthesia, followed by postoperative patient-controlled morphine analgesia (IV-PCA) for postoperative pain. Intra-operatively, hemodynamic changes indicative of pain will be treated with intravenous remifentanil (see below).

Group 2 will be administered with a continuous infusion of IV remifentanil supported by a single bolus of IV morphine, 0.2 mg/kg at the end of surgery, followed by IV-PCA morphine [15, 16].

Patients will be followed for three days post-operatively. The primary endpoint of this study is postoperative pain, which will be evaluated by several parameters:

1. A subjective visual analogue pain score (VAS, scale 0-10 cm) during rest, while coughing.
2. Time to first postoperative request of analgesia (from IV PCA).
3. Cumulative postoperative analgesia consumption (demand/delivery ratio).
4. Need for supplementary of alternative analgesia

The secondary endpoints will include levels of sedation, using the Wilson sedation score [17], length of time with indwelling urinary catheter, time to ambulation (sitting, walking), length of stay in the intensive care unit (ICU) and total length of hospitalization, time to extubation, need for re-intubation and analgesia-related adverse effects (see detailed patients' assessment).

Patient assessment All patients will be assessed in the first three postoperative days by the acute pain service during the morning hours (7-10am).

Primary endpoints

Pain control will be assessed according to the following measures:

* VAS [ranging from "0" (no pain) to "10" (worst imaginable pain)] in the morning (between 7-10am) and afternoon (between 13-15) on POD 1,2,3. Pain will be evaluated at rest and during coughing.
* The rate of IV-PCA activation (i.e., the number of times the delivery button was pressed) will be recorded daily (including within the lockout period), in order to evaluate both the demand and the consumption of postoperative analgesia, and document those patients whose analgesic needs were not fulfilled (with an activation-to-delivery rate ratio >1.5) [18].
* Cumulative morphine consumption will be assessed every 24 hours.
* The time of first request of postoperative analgesia and any need of extra boluses of analgesia or rescue drug (including dosages) will be recorded.

Secondary endpoints

Secondary outcome measures will include:

* Any opioid-related complications: respiratory depression (defined as hypoventilation, hypercapnia, and respiratory acidosis. Clinically manifested when PaCO2>60mmHg, and blood pH<7.25); nausea/vomiting; pruritus; sedation; allergic events.
* Any spinal-related complications will be recorded, e.g. postdural puncture headache.
* Intraoperative hemodynamic and/or respiratory complications; time to extubation.
* The time to ambulation (sitting, walking), and dependence on indwelling urinary catheter will be recorded..
* Sedation levels will be measured with the Wilson sedation scale (1, fully awake and oriented; 2,drowsy; 3, eyes closed, but rousable with command; 4, eyes closed, but rousable with mild physical stimulation; 5, eyes closed, not rousable with mild physical stimulation) will be recorded at times of pain assessment.
* Overall patients' satisfaction with pain relief will be evaluated with a 4-stage scale ("very good," "good," "moderate," or "bad") once daily, during afternoon visit.
* Additional data we will record include demographics (age, gender, weight, ASA), operative data (e.g. duration of surgery, amount of fluids and blood administered).

REFERENCES

1. Ballantyne, J.C., et al., Does the evidence support the use of spinal and epidural anesthesia for surgery? J Clin Anesth, 2005. 17(5): p. 382-91.
2. Cousins, M.J. and L.E. Mather, Intrathecal and epidural administration of opioids. Anesthesiology, 1984. 61(3): p. 276-310.
3. Kehlet, H. and K. Holte, Effect of postoperative analgesia on surgical outcome. Br J Anaesth, 2001. 87(1): p. 62-72.
4. Yeager, M.P., et al., Epidural anesthesia and analgesia in high-risk surgical patients. Anesthesiology, 1987. 66(6): p. 729-36.
5. Pelton, J.J., J.P. Hoffman, and B.L. Eisenberg, Comparison of liver function tests after hepatic lobectomy and hepatic wedge resection. Am Surg, 1998. 64(5): p. 408-14.
6. Vandermeulen, E.P., H. Van Aken, and J. Vermylen, Anticoagulants and spinal-epidural anesthesia. Anesth Analg, 1994. 79(6): p. 1165-77.
7. Matot, I., et al., Epidural anesthesia and analgesia in liver resection. Anesth Analg, 2002. 95(5): p. 1179-81, table of contents.
8. De Pietri, L., et al., The use of intrathecal morphine for postoperative pain relief after liver resection: a comparison with epidural analgesia. Anesth Analg, 2006. 102(4): p. 1157-63.
9. Redai, I., J. Emond, and T. Brentjens, Anesthetic considerations during liver surgery. Surg Clin North Am, 2004. 84(2): p. 401-11.
10. Sakowska, M., et al., A change in practice from epidural to intrathecal morphine analgesia for hepato-pancreato-biliary surgery. World J Surg, 2009. 33(9): p. 1802-8.
11. Milne, S.E., P.G. Horgan, and G.N. Kenny, Target-controlled infusions of propofol and remifentanil with closed-loop anaesthesia for hepatic resection. Anaesthesia, 2002. 57(1): p. 93.
12. Devys, J.M., et al., Intrathecal + PCA morphine improves analgesia during the first 24 hr after major abdominal surgery compared to PCA alone. Can J Anaesth, 2003. 50(4): p. 355-61.
13. Gwirtz, K.H., et al., The safety and efficacy of intrathecal opioid analgesia for acute postoperative pain: seven years' experience with 5969 surgical patients at Indiana University Hospital. Anesth Analg, 1999. 88(3): p. 599-604.
14. Swart, M., J. Sewell, and D. Thomas, Intrathecal morphine for caesarean section: an assessment of pain relief, satisfaction and side-effects. Anaesthesia, 1997. 52(4): p. 373-7.
15. Hansen, E.G., et al., Intra-operative remifentanil might influence pain levels in the immediate post-operative period after major abdominal surgery. Acta Anaesthesiol Scand, 2005. 49(10): p. 1464-70.
16. Schuttler, J., et al., A comparison of remifentanil and alfentanil in patients undergoing major abdominal surgery. Anaesthesia, 1997. 52(4): p. 307-17.
17. Wilson, E., et al., Sedation during spinal anaesthesia: comparison of propofol and midazolam. Br J Anaesth, 1990. 64(1): p. 48-52.
18. Weinbroum, A.A., et al., Dextromethorphan for the reduction of immediate and late postoperative pain and morphine consumption in orthopedic oncology patients: a randomized, placebo-controlled, double-blind study. Cancer, 2002. 95(5): p. 1164-70.

ELIGIBILITY:
Inclusion Criteria:

ASA physical status I-III patients (> 18 years old), scheduled for elective liver resection, pancreatic resection or pancreaticoduodenectomy ("Whipple" procedure) at Tel Aviv-Sourasky Medical Center.

Exclusion Criteria:

Contraindications to the spinal technique, allergy to the study drugs, patients treated with opioids for chronic pain, patients with obstructive sleep apnea, morbidly obese patients, pregnant women, patient requiring mechanical ventilation at the end of surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-11 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 72 hours
  Pain will be assessed 72 hours post-operatively by:
  1. A subjective visual analogue pain score (VAS, scale 0-10 cm) during rest, while coughing.
  2. Time to first postoperative request of analgesia (from IV PCA).
  3. Cumulative postoperative analgesia consumption (demand/delivery ratio).
  4. Need for supplementary of alternative analgesia

SECONDARY OUTCOMES:
Recovery and adverse effects | 72 hours
  Secondary outcomes will include: levels of sedation, length of time with indwelling urinary catheter, time to ambulation (sitting, walking), length of stay in the intensive care unit (ICU) and total length of hospitalization, time to extubation, need for re-intubation and analgesia-related adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, professor, Study Chair — Tel-Aviv Sourasky Medical Center; Elena Parladansky, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel